CLINICAL TRIAL: NCT00500708
Title: Identifying Markers That Predict Ventricular Arrhythmia Risk
Brief Title: Diagnostic Investigation of Sudden Cardiac Event Risk
Acronym: DISCERN
Status: Completed | Type: Observational
Sponsor: CardioDx (Industry)
Responsible Party: Sponsor
Other Study IDs: CDX_000003; DISCERN (Other: CardioDx)
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Arrhythmia; Cardiovascular Diseases; Heart Failure; CVD
Keywords: Heart failure; Implanted Cardioverter Defibrillator; Biological Markers; Molecular Genetics; Coronary Heart Disease; Gene Expression; GES; CVD; CHD; Precision Medicine; Genome-wide association study; Cardiovascular Disease; CAD; GWAS; DISCERN
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Failure; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, buffy coat, spun plasma, saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of the DISCERN study is to develop and validate a genomic diagnostic assay to identify patients at increased risk for lethal ventricular arrhythmias and sudden cardiac death (SCD).

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study. The research will be performed in three phases, each using distinct patient cohorts:

Phase I: Discovery - genes/biomarkers/clinical factors Phase II: Algorithm Development Phase III: Assay Validation

The final algorithm (Assay) may incorporate a combination of factors including genetic markers, biomarker(s), and clinical factor(s). Participation in the study does not alter clinical care. The procedures required by the protocol are collection of a research blood sample (at baseline only) and interviews with the subject to collect specific clinical information at baseline and follow-up (6 mos, 1 yr, 2 yr, 3 yr, 4 yr, and 5 yr) after enrollment. All other data collected is in accordance with the participating institution's standard patient care.

ELIGIBILITY:
Inclusion Criteria:

* Implantable cardiac defibrilIator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) implanted for primary prevention
* Left ventricular ejection fraction (LVEF) ≤ 50 %
* Ability to collect clinical follow-up and endpoint information, including device interrogation data

Exclusion Criteria:

* Congenital heart disease
* Known inherited arrhythmia disorder
* Organ transplantation
* Inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's with ventricular dysfunction (low ejection fraction) undergoing implantation of ICD or CRT-D for primary prevention. Patient's may be enrolled at time of implant or during follow-up in electrophysiology clinic as long as full device records are available since time of implant.
Sampling Method: Probability Sample
Enrollment: 1564 (Actual)
Dates: Start 2007-07; Primary Completion 2011-08-01 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
Gene discovery | up to 3 years
  Genome Wide Association Study (GWAS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, Study Director — CardioDx, Inc.
Locations (8):
- United States (8):
  - Alaska Heart Institute, Anchorage, Alaska
  - Palo Alto Medical Foundation, Palo Alto, California
  - Minneapolis Heart Institute and Foundation, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - West Penn Allegheny Health System, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Healthcare, Salt Lake City, Utah

REFERENCES:
- [Result] Hranitzky PM, Sehnert AJ, Blanchard JL, et al. Abstract 16410: Identification of novel genetic markers associated with lethal ventricular arrhythmias in heart failure patients: genome wide association study in the DISCERN cohort. Circulation. 2010;122. Abstract 16410.